CLINICAL TRIAL: NCT03803293
Title: Right Drug, Right Dose, Right Time - Using Genomic Data to Individualize Treatment (The RIGHT Protocol)
Brief Title: Right Drug, Right Dose, Right Time - Using Genomic Data to Individualize Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Suzette J. Bielinski, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12-003371
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects
Keywords: Pharmacogenomics; Personalized Medicine; Pharmacogenomic Varients
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: The Mayo Clinic Biobank is an institutional resource comprised of adult community volunteers who donated biological specimens, provided risk factor data, access to EHR data, and consented to participate in additional studies. Subjects in the Mayo Clinic Biobank are the cohort that was recruited to participate in the RIGHT study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary cohort (Other): All eligible Biobank participants that receive the majority of their care at Mayo Clinic based on EHR length and depth had pharmacogenomic testing done.
  Interventions: Diagnostic Test: Pharmacogenomic testing

INTERVENTIONS:
Diagnostic Test: Pharmacogenomic testing — A comprehensive PGx interpretive report created by OneOme (www.oneome.com) provides information on how an individual patient's genes may affect medication response. OneOme utilizes algorithms and curated clinical PGx knowledge to generate a highly intuitive personalized report based on a patient's genomic results.

SUMMARY:
This study is being done to better understand how genetic information related to drug dosing and use can affect medical care of patients. By doing this study, the investigators are developing and improving ways to incorporate information about drug related genetic variants into the medical record.

DETAILED DESCRIPTION:
The purpose of this research is to initiate a test of the concept that sequence information can be coupled to electronic medical records (EMRs) for use in healthcare.The focus of this study is on pharmacogenomics, given the role of adverse drug reactions (ADRs) as major causes of morbidity and mortality, the increasing number of recognized variants included in FDA labels as mediators of both efficacy and toxicity, and the relative lack of stigma attached to carriers of variants in "pharmacogenes". Preemptive sequencing of patients interrogates large numbers of PGx variants and integrates clinically actionable results in a patient's electronic health record (EHR) for use by clinicians at the point-of-care. It is unknown, however, whether integration of preemptive PGx data into the EHR will significantly improve patient outcomes and reduce healthcare costs. Therefore, the Right Drug, Right Dose, Right Time Using Genomic Data to Individualize Treatment Protocol (RIGHT Protocol) study was designed to recruit a large group of patients for preemptive PGx testing, to develop the EHR infrastructure to deliver clinical decision support in real time, and to study the effects of integrating preemptive PGx testing into clinical practice on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Biobank participants who receive the majority of their care at Mayo Clinic based on EHR length and depth.

Exclusion Criteria:

* Not in the Mayo Clinic Biobank. Do not receive the majority of their care at a Mayo Clinic site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11098 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Study Participants - Total number of subjects identified with high risk for being prescribed a PGx drug | Baseline
  Total number of subjects identified with high risk for being prescribed a PGx drug

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Bielinski, PhD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials